CLINICAL TRIAL: NCT02378792
Title: The Clinical Research on TsingHua Vagus Nerve Stimualtor for Treatment of Refractory Epilepsy
Brief Title: Clinical Trial of Vagus Nerve Stimulation for Treatment of Refractory Epilepsy
Acronym: VNSRE
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Pins Medical Co., Ltd (Industry)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PINS-012
Record Dates: First submitted 2015-02-27; First posted 2015-03-04 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-04

CONDITIONS: Refractory Epilepsy
Keywords: PINS VNS Refractory Epilepsy
MeSH Terms: conditions — Drug Resistant Epilepsy | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vagus Verve Stimulation is on (Experimental)
  Interventions: Device: Vagus Nerve Stimulation
- Placebo Vagus Verve Stimulation is off (Sham Comparator)
  Interventions: Device: Vagus Nerve Stimulation

INTERVENTIONS:
Device: Vagus Nerve Stimulation — Vagus Nerve Stimulator
  Other Names: PINS Stimulator System

SUMMARY:
Evaluate the long-term clinical effectiveness and safety of the PINS vagus nerve stimulator to patients with refractory epilepsy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 6-60.
2. Having tried at least two appropriate anti-epileptic drugs (AEDs) tested to tolerance or to blood levels at upper end of the target range of which at least 2 have been tolerated at normal dose.
3. At least 1 seizure per month.
4. In good health except epilepsy.
5. With normal MMSE score
6. Patients or his(her) familyscould understand this method and sign the informed consent 7）Patients with good compliance and could complete postoperative follow-up.

Exclusion Criteria:

1. Results of MRI remind epilepsy caused by intracranial space-occupying lesions.
2. The vagus nerve lesion and damage
3. Tumor, cardiopulmonary anomaly, progressive neurological diseases, asthma，mental disease，pepticulcer，diabetes Type 1，bad health etc, and other surgical contraindication
4. Alcohol addiction, smoking, and sleep-related breathing disorders

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-08; Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Changes in seizure frequency from baseline to the seizure count evaluvation period 6 month | 4,8,12,16,20,24 months of stimulation

SECONDARY OUTCOMES:
Changes in seizure frequency from baseline to the seizure count evaluvation period | 4,8,12,16,20,24 months of stimulation
  Changes in seizure frequency from baseline to 4,8,12,16,20,24 months
Overall Quality of Life in Epilepsy-31 (QOLIE-31) Score in Patients With Baseline & at Least One Post-baseline QOLIE Assessment | Mean change from baseline QOLIE-31 Overall Score at 12,24 months
  QOLIE-31 contains 7 multi-item scales that tap the following health concepts:overall quality of life, emotional well-being, social functioning, energy/fatigue, worry about seizure,cognitive functioning,medication effects. Range of values 0-100. Higher scores reflect better quality of life; lower ones, worse quality of life.
Changes in the Number of Anti-epileptic Drugs Prescribed | At12,24 months
  Changes in Anti-Epileptic Drugs (AEDs) in patients with less then a 50% reduction in seizures
Changes from Basline in the Engel and McHugh description | At 12,24 months
Changes from Basline in 24 hour ECG description | At 12,24 months

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Beijing Tiantan Hospital, Beijing, Beijing Municipality
  - The first hospital of jilin university, Changchun, Jilin
  - The general of shenyang military, Shenyang, Liaoning
  - Qilu hospital of shandong university, Jinan, Shandong
  - The second affiliated hospital zhejiang university school of medicine, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Liu H, Zhan P, Meng F, Wang W. Chronic vagus nerve stimulation for drug-resistant epilepsy may influence fasting blood glucose concentration. Biomed Eng Online. 2020 May 29;19(1):40. doi: 10.1186/s12938-020-00784-1. PMID 32471438